CLINICAL TRIAL: NCT06621342
Title: Evaluating Cytokine Concentrations in the Endometrium Before and After Autologous Platelet Rich Plasma Uterine Infusion Preceding Frozen Embryo Transfer
Brief Title: Platelet Rich Plasma Uterine Infusion
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study deferred/stopped by initiator before any study recruitment was initiated.
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY00149149
Record Dates: First submitted 2023-01-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-01

CONDITIONS: Infertility; Endometriosis
Keywords: implantation failure; IVF; Embryo Transfer
MeSH Terms: conditions — Infertility; Endometriosis

STUDY DESIGN:
Intervention Model Description: 40 patients will be enrolled in each of the control and test groups, using a confidence interval of 95% and a 5% margin of error Total participants expected = 80.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: 2. It is not possible to blind clinical staff for the procedure. It is not necessary for the integrity of the study to blind participants as we are assessing their pregnancy outcomes. Regardless of which group they are assigned, participants will partake in routine prenatal care, as well as two additional study visits. They will know which group they have been assigned at the time of the procedure based on if they receive the treatment prior to implantation or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP Experimental (Experimental): The treatment group will receive 1 ml of autologous PRP infused into the cervix via Rocket IUI catheter at 72+/- 5 hours and 48 +/- 5 hours prior to embryo transfer. Prior to the first PRP infusion, endometrial secretions will be aspirated as described in a previous study regarding endometrial secretions. An embryo transfer catheter will be introduced trans-cervically. A 2 mL syringe will be used to gradually add suction, aspirating secretions from the endometrium. The outer sheath of the embryo catheter will be positioned in the exterior, and the inner catheter retracted into the outer sheath, to avoid cervical fluid contamination in the collected endometrial secretions. Secretions will be deposited into screw top cryovials by snipping the end of the transfer catheter containing secretion off into the tube. These tubes will then be snap-frozen in liquid nitrogen. Process will be repeated prior to embryo transfer
  Interventions: Biological: PRP Experimental
- PRP Control (Placebo Comparator): Negative control patients will have endometrial secretions aspirated at identical intervals to the test group but will not receive PRP infusions.
  Interventions: Biological: PRP Experimental

INTERVENTIONS:
Biological: PRP Experimental — All participants will have 5 2ml tubes of blood collected at 72 +/- 5 hr prior to embryo transfer and again at 48 +/- 5 hour prior to embryo transfer. This blood will be processed to create PRP for the uterine infusion per protocol.

SUMMARY:
Platelet Rich Plasma (PRP), a rich source of important growth factors, has been shown to significantly affect the body's ability to heal and regenerate tissues. It is an affordable, accessible treatment with little risk of side effects that is being utilized in many areas of regenerative and cosmetic medicine. PRP is also relatively easy to prepare with supplies on hand in most IVF clinics. Specifically relating to reproductive function, PRP has been demonstrated to increase cellular proliferation and decrease fibrosis in damaged rat endometrium. It is hypothesized that infusing the uterus with Platelet Rich Plasma at measured intervals prior to embryo transfer will increase concentrations of implantation-promoting cytokines while reducing concentrations of inflammatory cytokines during the window of implantation.

DETAILED DESCRIPTION:
1. Platelet Rich Plasma (PRP), a rich source of important growth factors, has been shown to significantly affect the body's ability to heal and regenerate tissues.7 It is an affordable, accessible treatment with little risk of side effects that is being utilized in many areas of regenerative and cosmetic medicine. PRP is also relatively easy to prepare with supplies on hand in most IVF clinics. PRP has shown great promise in veterinary medicine to regenerate tissues and reduce endometrial inflammation.8 Specifically relating to reproductive function, PRP has been demonstrated to increase cellular proliferation and decrease fibrosis in damaged rat endometrium.6 Endometritis, which is characterized by an increase in inflammatory cells, erosion of the endometrial epithelial layer as well as endometrial edema has been a large cause of infertility in cattle and therefore revenue loss in the cattle industry. A recent study applying uterine infusion of PRP as the intervention demonstrated decreased markers for inflammation in cattle in vivo and as well as decreased inflammatory markers in in vitro cultured endometrial cells exposed to PRP.6 A similar in vitro study was conducted on horses; the authors noticed a decrease in clinical uterine infections in mares along with an increased embryo recovery rate.31 Chronic endometritis is hypothesized to be one of the potential factors involved in recurrent implantation failure in women.32 Using these previous studies in veterinary medicine as a model for potential benefit in human patients, it would be prudent to explore the mechanism of PRP action in humans. It is hypothesized that infusing the uterus with Platelet Rich Plasma at measured intervals prior to embryo transfer will increase concentrations of implantation-promoting cytokines while reducing concentrations of inflammatory cytokines during the window of implantation. TGF-b, IL-6 and LIF are known to be promoters of implantation, while TNF-a and IL-4 are pro-inflammatory factors and can inhibit implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient at REI clinic population
* Ages 23 to 45
* Undergo frozen embryo transfers with clinic standard medicated protocols
* Transferring one or two embryos on day 5 or 6 of development

Exclusion Criteria:

* BMI >32
* Low level or high-level mosaic
* Aneuploid embryos only will be excluded
* Desiring day 3 or fresh embryo

Ages: 23 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients assigned female at birth, who are capable of becoming pregnant.
Enrollment: 0 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Determine the effect of autologous uterine PRP infusion on factors critical to the implantation process | 18 months
  Compare differences of the levels TGF- b, IL-6 and LIF in endometrial secretions pre- and post-treatment.

SECONDARY OUTCOMES:
Determine the effect of autologous uterine PRP infusions on factors that are deleterious to embryo implantation | 18 months
  By measuring and comparing levels of TNF-a and IL-4 post uterine infusion with PRP.

OTHER OUTCOMES:
Determine if autologous uterine PRP infusion influences implantation rates after frozen embryo transfer. | 18 months
  Compare implantation rates after frozen embryo transfer post PRP infusion to implantation rates in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Marsh, MD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No